CLINICAL TRIAL: NCT03406000
Title: A 28-week, Prospective, Single-arm, Phase 4 Study to Evaluate Treatment Optimization With Once-daily Insulin Glargine 300 U/mL in Combination With Prandial Rapid-acting Insulin Analogue in Patients With Type 1 Diabetes Previously Uncontrolled on Twice-daily Basal Insulin as Part of Basal-bolus Therapy
Brief Title: Phase 4 Study to Evaluate Treatment Optimization With Once-daily Insulin Glargine 300 U/mL
Acronym: TOP1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLARGL08200; U1111-1186-2485 (Other: UTN)
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Type I Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insulin glargine (U300) (Experimental): Self-administered subcutaneously once daily in the morning, at the same time.The initial dose for patients switching from insulin glargine is 80% of the total daily dose of basal insulin agent that was discontinued. Thereafter, insulin glargine (U300) will follow a titration algorithm for dose adjustment.
  Interventions: Drug: INSULIN GLARGINE (U300)

INTERVENTIONS:
Drug: INSULIN GLARGINE (U300) — Pharmaceutical form: Solution for Injection
  Route of administration: Subcutaneous injection
  Other Names: Toujeo, HOE901

SUMMARY:
Primary Objective:

To evaluate the efficacy of switching treatment from twice-daily basal insulin to once-daily insulin glargine (U300) as part of basal bolus regime in terms of glycated hemoglobin improvement (reduction by at least 0.3%), in uncontrolled type 1 diabetes mellitus patients.

Secondary Objectives:

* To evaluate other efficacy parameters in terms of glycemic control as well as safety including hypoglycemia events, weight changes, and adverse events.
* To evaluate the effect of insulin glargine (U300) on diabetes treatment satisfaction and fear of hypoglycemia as well as patient's satisfaction regarding the number of daily injections.

DETAILED DESCRIPTION:
The estimated average study duration is 29 weeks, including run-in period of 4 weeks; treatment period of 24 weeks, and follow-up period of 1 week.

ELIGIBILITY:
Inclusion criteria :

* Male or Female.
* Age ≥ 18 years.
* With Type 1 diabetes mellitus.
* Being treated twice-daily with any basal insulin in combination with prandial rapid-acting insulin analogue for at least one year.
* Have an glycated hemoglobin (HbA1c) measurement of 7.5% - 10.0% at study entry.
* Patients who have signed an Informed Consent Form.

Exclusion criteria:

* Type 2 diabetes mellitus.
* Known hypoglycemia unawareness
* Repeated episodes of severe hypoglycemia or diabetes ketoacidosis within the last 12 months.
* End-stage renal failure or being on hemodialysis.
* Any clinically significant abnormality identified on physical examination, laboratory tests, or vital signs at the time of screening or baseline, or any major systemic disease resulting in short life expectancy that in the opinion of the Investigator would restrict or limit the patient's successful participation for the duration of the study.
* Known hypersensitivity / intolerance to insulin glargine or any of its excipients.
* Patients treated with glucagon like peptide agonists.
* Use of systemic glucocorticoids (excluding topical application or inhaled forms) for one week or more within 90 days prior to the time of screening.
* Pregnant or lactating women.
* Women of childbearing potential with no effective contraceptive method.
* Participation in another clinical trial.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

PRIMARY OUTCOMES:
Mean change in HbA1c | From baseline to Week 24
  Mean change in glycated hemoglobin (HbA1c) from baseline to Week 24 (%)

SECONDARY OUTCOMES:
Mean change in HbA1c | From baseline to Week 12
  Mean HbA1c change from baseline to Week 12
Mean change in fasting plasma glucose (FPG) | From baseline to Week 12 and Week 24
  Mean change in FPG from baseline to Week 12 and Week 24
Mean change in fasting SMBG | From baseline to Week 12 and Week 24
  Mean change in fasting self-monitored blood glucose (SMBG) from baseline to Week 12 and Week 24
Mean change in 8-point SMBG | From baseline to Week 12 and Week 24
  Mean change in 8-point SMBG from baseline to Week 12 and Week 24
Proportion of patients achieving HbA1c target of <7.0% | At Weeks 12 and 24
  Proportion of patients achieving HbA1c target of <7.0% at Week 12 and Week 24
Proportion of patients achieving HbA1c target of <7.0% without hypoglycemia event | At Weeks 12 and 24
  Proportion of patients achieving HbA1c target of <7.0% without hypoglycemia event during the last 4 weeks of treatment
Proportion of patients achieving HbA1c improvement of at least 0.3% without nocturnal hypoglycemia | From baseline to Week 24
  Proportion of patients achieving HbA1c improvement from baseline to week 24 of at least 0.3% without nocturnal hypoglycemia (documented <70 mg/dL) and/or severe hypoglycemia (between 00.00 and 05:59 am SMBG) during the last 4 weeks of treatment
Proportion of patients with any improvement in HbA1c | From baseline to Week 24
  Proportion of patients with any improvement in HbA1c from baseline to week 24 and decrease in occurrence of nocturnal hypoglycemia (nocturnal defined as time between 00.00 and 05:59 am) evaluated from baseline to Week 24
Proportion of patients with no deterioration in HbA1c | From baseline to Week 24
  Proportion of patients with no deterioration in HbA1c from baseline to week 24 and decrease in occurrence of nocturnal hypoglycemia
Proportion of patients with no deterioration in HbA1c | From baseline to Week 24
  Proportion of patients with no deterioration in HbA1c from baseline to week 24 and no increase in occurrence of nocturnal hypoglycemia
Adverse events (AEs) | Up to 28 weeks
  Number of adverse events and serious adverse events
Mean change in body weight | From baseline to Week 12 and Week 24
  Mean change in body weight from baseline to Weeks 12 and 24
Mean change in daily insulin doses | From baseline to Week 24
  Insulin glargine (U300) dose: Mean change in daily insulin doses (basal, prandial, total) from baseline to Week 24
Number of patients experiencing hypoglycemia | Up to 28 weeks
Proportion of patients experiencing hypoglycemia | Up to 28 weeks
Number of hypoglycemic events per patient-year | Up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (11):
- Brazil (11):
  - Investigational Site Number 076013, Campinas
  - Investigational Site Number 076016, Curitiba
  - Investigational Site Number 076007, Curitiba
  - Investigational Site Number 076005, Fortaleza
  - Investigational Site Number 076002, Goiânia
  - Investigational Site Number 076004, Porto Alegre
  - Investigational Site Number 076011, Ribeirão Preto
  - Investigational Site Number 076006, São José dos Campos
  - Investigational Site Number 076015, São Paulo
  - Investigational Site Number 076012, São Paulo
  - Investigational Site Number 076001, São Paulo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Dualib PM, Dib SA, Augusto GA, Truzzi AC, de Paula MA, Rea RR. Effect of switching from twice-daily basal insulin to once-daily insulin glargine 300 U/mL (Gla-300) in Brazilian people with type 1 diabetes. Diabetol Metab Syndr. 2024 Jul 9;16(1):152. doi: 10.1186/s13098-024-01385-x. PMID 38982528